CLINICAL TRIAL: NCT04583917
Title: Brain INvolvement in Dystrophinopathies (BIND): Deep Functional Phenotyping of Duchenne Muscular Dystrophy and Becker Muscular Dystrophy Patients (WP5) Part 1: a Multicentre Online Phenotyping and Neurobehavioural Data Collection Study
Brief Title: Brain Involvement in Dystrophinopathies Part 1
Status: Completed | Type: Observational
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other); Leiden University Medical Center (Other); Stichting Kempenhaeghe (Unknown); Region Hovedstadens Apotek (Other Government); Institut Necker Enfants Malades (Other); Catholic University of the Sacred Heart (Other); Università degli Studi di Ferrara (Other); Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Other Study IDs: 20NM34
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Duchenne Muscular Dystrophy; Becker Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to collect data from a large cohort of individuals with DMD and BMD focusing on the neurobehavioural aspects of these conditions and their correlation to the location of the DMD gene mutation.

DETAILED DESCRIPTION:
Intellectual disability and neurobehavioural comorbidities affect at least 50% of the individuals with Duchenne muscular dystrophy (DMD), which, although a rare genetic disease, is the most common form of muscular dystrophy in childhood. Several studies have documented that 25% of the DMD population has intellectual disability with recent studies suggesting that autism and clinically relevant hyperactivity affects 20% and 25% of DMD boys respectively. A milder allelic variant, named Becker muscular dystrophy (BMD), has similar prevalence in the population and is also associated with variable degrees of central nervous system (CNS) comorbidities, which however have been less well defined.

The investigators will address these deficiencies in a large multicentre study funded by the European Commission (EU H2020) involving 6 countries (Denmark; The Netherlands; France; Spain; Italy and UK) with the largest European neuromuscular centres and advocacy groups. The aim will be to study the neurobehavioural aspects of DMD and BMD as well as their correlation to the genotype. This study will involve male participants with DMD aged 5-17 years and with BMD aged 5-50 years. It will comprise of online questionnaires that will be completed either by a parent of a participant <17 years or an adult participant. The questionnaires take approximately 70 minutes to complete, however this can be done in multiple sittings. Currently there is a lack of information to assist the prognosis of CNS comorbidities, as existing databases and registries typically focus on the motor milestones and physical disability of these patients. There is therefore, an urgent need to present the course and outcomes in DMD and BMD patients with a wide range of DMD mutations, to provide information at the point of diagnosis and onwards for families, clinicians and service providers. It will also assist in paving the way to greater biological understanding and personalization of interventions.

ELIGIBILITY:
Inclusion Criteria:

For DMD patients:

* Male
* age 5-17 years
* genetically-proven diagnosis of DMD
* genetic mutation that abrogates expression of Dp427 alone (assigned in DMD Group 1: Dp427-/Dp140+) or both Dp427 and Dp140 (assigned to DMD Group 2: Dp427-/Dp140-); or all isoforms (assigned to DMD group 3)

For BMD patients:

* age 5-50 years
* genetically-proven diagnosis of BMD
* genetic mutation that decreases expression of Dp427 alone (assigned to BMD Group 1), of both Dp427 and Dp140 (assigned to BMD Group 2), or of all the isoforms (assigned to BMD group 3).

Exclusion Criteria:

* Lack of a molecular diagnosis of DMD or BMD
* Mutation falls outside the regions of interest
* A severe co-morbidity or planned surgical intervention within 6 months from the study which could interfere with the well-being of the participant

Ages: 5 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — DMD and BMD are sex-linked conditions, which occur predominantly in males.
Study Population: Patients will be those followed in the two neuromuscular centres located in London and Newcastle; via the UK Clinical North Star network, the BIND website and the UK advocacy groups MDUK, Action Duchenne and Duchenne UK. A similar recruitment process will take place in the other EU countries, according to local regulations and after having obtained the relevant local ethical approval.
Sampling Method: Non-Probability Sample
Enrollment: 377 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
CNS Comorbidity Pheotyping | 90 minutes
  Correlate CNS comorbidity phenotypes with genotype in DMD and BMD patients

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Muntoni, Principal Investigator — University College, London
Locations (7):
- Copenhagen Neuromuscular Center, Copenhagen, Denmark
- Imagine Institut Des Maladies Genetiques Necker Enfants Malades Fondation, Paris, France
- Universita Cattolica Del Sacro Cuore, Rome, Italy
- Stichting Kempenhaeghe, Heeze, Netherlands
- Universidad Complutense de Madrid, Madrid, Spain
- United Kingdom (2):
  - GOSH/UCL, London
  - University of Newcastle Upon Tyne, Newcastle

IPD SHARING:
Plan to Share IPD: Undecided
Pseudonymised data will be shared amongst collaborating partners in the project, but details on data sharing are still under discussion.

REFERENCES:
- See also: BIND: Brain Involvement in Dstrophinopathies study website — https://bindproject.eu/